CLINICAL TRIAL: NCT00627900
Title: Model Project for the Reduction of Coronary Restenosis
Brief Title: Cost-Effectiveness Study in the Reduction of Coronary Restenosis With Sirolimus-Eluting Stents
Acronym: GERSHWIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Techniker Krankenkasse (Other)
Responsible Party: Frau Jena Benkenstein, Techniker Krankenkasse
Allocation: Non-Randomized
Other Study IDs: EK-Vorgang: Verschiedenes
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS (Other): Implantation of a bare metal stent
  Interventions: Device: bare metal stent
- SES (Other): Implantation of a sirolimus-eluting stent
  Interventions: Device: Cypher-Stent (Implantation of a sirolimus-eluting stent)

INTERVENTIONS:
Device: bare metal stent — implantation of a bare metal stent
  Arms: BMS
Device: Cypher-Stent (Implantation of a sirolimus-eluting stent) — Implantation of a sirolimus-eluting stent
  Other Names: Cypher-Stent
  Arms: SES

SUMMARY:
Since the advent of coronary stents, in-stent restenosis has proven to be the major limitation of interventional cardiology, occurring in as many as 30% of patients. Drug-eluting stents are specifically designed to prevent the problem of in-stent restenosis. They consist of a selective anti-proliferative drug, sirolimus, a controlled-release polymer, and a closed-cell stent delivery platform. Upon placement, sirolimus elutes into the vessel wall and stops the process of neointimal hyperplasia, thereby significantly reducing the incidence of in-stent restenosis.

The study "Prevention of Coronary Restenosis" examines the effectiveness of sirolimus-eluting stents (SES) compared to bare-metal stents (BMS) in patients with coronary stenosis. The goal of the study is to examine whether the guideline-supported implantation of SES, despite the higher initial cost, improves the quality and economic outcomes of the treatment of patients with coronary stenosis. Secondarily, the study evaluates patient quality of life, impairment of daily activities, re-intervention rate, as well as an account of the utilisation and benefits of the implemented standardised guidelines.

In this prospective, multi-centre, country-wide cohort study, 658 patients undergoing an implantation of a SES for treatment of coronary stenosis were recruited from 35 hospital centres. Their treatment and outcomes will be evaluated over a 3-year period by means of standardised questionnaires. In addition, information obtained from the patients will be confirmed and augmented by telephone interviews with the attending physicians involved in their follow-up care.

In order to appraise the effect of the new therapy, a comparison cohort group of 394 patients receiving a BMS was recruited. These patients will be evaluated and observed by the same method as those patients receiving a drug-eluting stent, also over 3 years

ELIGIBILITY:
Inclusion Criteria:

* indication for implantation of a coronary stent
* de novo lesions < or = 30 mm in patients with diabetes
* de novo lesions 12-30 mm or RVD 2.5-3.00 mm in patients without diabetes

Exclusion Criteria:

* acute MI
* lesion length >30 mm
* in-stent restenosis
* distal lesion in RVD < 2.25 mm
* lesion in left main or bypass vessel
* contraindication to Clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2003-04; Primary Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Cost equivalence of sirolimus-eluting coronary stents versus bare metal stents | 3,6,12,18,24, 36 months following stent implantation

SECONDARY OUTCOMES:
MACE (re-PCI, myocardial infarction, CABG, death) | 3,6,12,24,36 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, MD, MPH, MBA, Study Director — Charite University, Berlin, Germany
Locations (1):
- Institut für Sozialmedizin, Epidemiologie und Gesundheitsökonomie, Berlin, Germany

REFERENCES:
- [Result] Bruggenjurgen B, McBride D, Bode C, Hamm CW, Kuck KH, Willich SN. Sirolimus-eluting versus bare-metal stents for the reduction of coronary restenosis: 18-month angiographic results from the GERSHWIN Study. Herz. 2007 Dec;32(8):650-5. doi: 10.1007/s00059-007-3048-2. PMID 18060612